CLINICAL TRIAL: NCT03732261
Title: Effects of Exercise and Yogurt on Bone Mineral Density and Immunological Factors in Human Milk: The MEEMA Study
Acronym: MEEMA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID 19 pandemic
Sponsor: North Carolina Agriculture & Technical State University (Other)
Responsible Party: Principal Investigator, Heather Colleran, Assistant Professor, North Carolina Agriculture & Technical State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MEEMA
Record Dates: First submitted 2018-10-19; First posted 2018-11-06 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Lactational Amenorrhea; Body Weight Changes; Bone Loss
Keywords: postpartum, lactation, bone density, exercise, yogurt
MeSH Terms: conditions — Body Weight Changes; Bone Diseases, Metabolic; Breast Feeding; Motor Activity | interventions — Exercise; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention Group: Women randomized to the intervention group will be given a 3month membership to a community based exercise program, a pedometer and individual dietary recommendations. They will be asked to attend a minimum of three 45 minute to 60 minute exercise sessions per week but no more than five and will gradually build to walk 10,000 steps per day. Childcare and breastfeeding support will be provided. Trained research assistants will lead all group sessions. Weekly workout volume will be calculated and weekly steps will be monitored by research assistants. For the dietary intervention, the women will be provided 6oz of plain yogurt fortified with vitamin D post workout for the 12-week intervention. If any yogurt is out of date (expired), we will dispose of the expired yogurt. Weekly monitoring for the consumption of the yogurt and energy intake will be conducted by face-to-face or telephone interviews by research assistants.
  Interventions: Other: Exercise and dietary
- Control (No Intervention): Minimal Care Group: Women randomized into the minimal care group will be asked not to participate in any structured exercise or make any changes in their diet. They will be permitted to walk their infants in strollers at a leisurely pace (no faster than 2 mph) for no more than 30 minutes per day. After the endpoint measurements of the 12-wk intervention, the minimal care group will be asked to join the community based program provided to the intervention group. The participants will be given the pedometer, individual dietary recommendations and yogurt. Additionally, support by the PI and research assistants for exercise and diet will be provided until the one-year postpartum laboratory measurement.

INTERVENTIONS:
Other: Exercise and dietary — The 12-week study invention will take place between 6 to 8-weeks postpartum and 18 to 20-weeks postpartum, with a follow-up at one year postpartum. The six-week postpartum time point is to allow for exercise clearance from the participant's obstetrician. The exercise clearance is needed prior to the baseline laboratory measurement. Women will be randomized to an intervention group or minimal care group after all baseline measurements (anthropometrics, cardiovascular fitness test, human milk and blood samples and DXA) at six-weeks postpartum. A random numbers table will be used to stratify by parity and determine groups.
  Arms: Intervention

SUMMARY:
Obesity in America has risen to epidemic levels over the past 20 years. For women, childbearing itself could be a contributing factor to this high prevalence of excess weight. In addition, for women who breastfeed, lactation is a time of rapid bone loss due to hyperprolactinemia, amenorrhea, and increased bone turnover, especially in the lumbar spine and hip. The American Academy of Pediatrics recommends exclusive breastfeeding for the first 6 months, continue to at least 12 months with the introduction of complementary foods and up to 2 years. Breastfeeding helps reduce long term maternal weight retention from pregnancy, the risk of childhood obesity and provides a number of immunological factors to promote the immune system and gastrointestinal system of the neonate.

Bone loss due to lactation is usually reversed with weaning; however, not all women recover from this bone loss which increases the risk of osteoporosis later in life. Weight bearing exercise and dairy intake (milk, yogurt, cheese) plus vitamin D supplementation may provide some protection from bone loss. Thus, the objective of this study is to promote long-term lifestyle changes that support healthy lifelong weight management through a community based exercise intervention and daily yogurt consumption program aimed at overweight- to- obese lactating postpartum women.

DETAILED DESCRIPTION:
The specific aims of this project are to evaluate in overweight lactating women at 6 and 20 weeks postpartum (PP) whether an exercise and yogurt supplementation intervention, compared to a minimal care group, will:

1. Improve body composition. The working hypothesis for this aim, based on previous studies (Lovelady et al 2009; Colleran et al 2012), is thatthe intervention group will have less loss of lean body mass and bone mineral density but more fat loss compared to the minimal care group at 20 weeks PP.
2. Promote an increase in cardiovascular fitness. The working hypothesis for this aim, based on previous studies (Lovelady et al 2009; Colleran et al 2012), is that the intervention group will exhibit an increase in predicted maximal oxygen consumption and maximal strength compared to the minimal care group at 20 weeks PP.
3. Increase immunological factors within breastmilk. The working hypothesis for this aim, based on a previous study (Lovelady et al 2003), is that the intervention group will exhibit an increase in IgA, lactoferrin, lysozyme and Bidfidus factor concentrations in breast milk which will improve immunological benefits to the nursing infant.

ELIGIBILITY:
Inclusion Criteria:

* women must be at least 2 weeks postpartum
* be between the ages of 25 to 40
* have a self-reported body mass index (BMI) between 25 and 35 kg/m2
* be fully breastfeeding (< 4 oz of formula given to the infant only on occasion)
* be sedentary for the past 3 months (< 3 weekly sessions of moderate aerobic activity)
* be non-smokers
* had a singleton birth.

Exclusion Criteria:

* delivery by cesarean section
* have medical complications where exercise was contraindicated
* have an inability to consume yogurt (i.e. maternal or infant allergies/intolerance to the dairy protein or sugar) or
* a have diagnosis with a disease that affects hormone levels.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Body composition: Bone Mineral Density | 12 weeks
  The working hypothesis for this aim, based on previous studies (Lovelady et al 2009; Colleran et al 2012), is that the intervention group will have less loss of lean body mass and bone mineral density but more fat loss compared to the minimal care group at 20 weeks PP.
Increase immunological factors within breastmilk | 12 weeks
  The working hypothesis for this aim, based on a previous study (Lovelady et al 2003), is that the intervention group will exhibit an increase in IgA, lactoferrin, lysozyme and Bidfidus factor concentrations in breast milk which will improve immunological benefits to the nursing infant.

SECONDARY OUTCOMES:
Cardiovascular fitness | 12 weeks
  The working hypothesis for this aim, based on previous studies (Lovelady et al 2009; Colleran et al 2012), is that the intervention group will exhibit an increase in predicted maximal oxygen consumption and maximal strength compared to the minimal care group at 20 weeks PP.

CONTACTS AND LOCATIONS:
Overall Officials: Heather L Colleran, PHD, Principal Investigator — North Carolina Agriculture & Technical State University
Locations (1):
- North Carolina A&T State University, Greensboro, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No